CLINICAL TRIAL: NCT00304720
Title: Tacrolimus and Mycophenolate Mofetil as Post-Grafting Immunosuppression After Conditioning With Fludarabine and Low-Dose Total Body Irradiation for Recipients of HLA-Matched Family Donor Hematopoietic Cell Transplants
Brief Title: Tacrolimus and MMF as Post Grafting Immunosuppression After Conditioning With Flu TBI for HLA Matched Family Donor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colorado Blood Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMBMT-124-A
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2004-03

CONDITIONS: Multiple Myeloma; Lymphoma; Acute Myelogenous Leukemia; Acute Lymphocytic Leukemia; Myelodysplastic Syndrome
Keywords: Lymphoma; Leukemia
MeSH Terms: conditions — Multiple Myeloma; Lymphoma; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia | interventions — Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus and MMF

SUMMARY:
Primary Objective:

A. To determine whether stable allogeneic hematopoietic engraftment can be safely established in patients receiving a non-myeloablative allogeneic SCT from a matched sibling donor, with fludarabine and low-dose TBI, with pre- and post-transplant immunosuppression with tacrolimus and MMF.

B. To evaluate the incidence of grade II-IV GVHD associated with this treatment.

DETAILED DESCRIPTION:
Conditioning regimen:

1. Days - 4 to -2: Fludarabine 30 mg/m2/day IV.
2. Day 0: TBI 2.0 Gy at 6-7 cGy/min from a linear accelerator, followed by stem-cell infusion. TBI will preferably be administered between 7:00 a.m. and 1:00 p.m. to avoid proximity to tacrolimus/MMF administration.

Immunosuppression:

Day -3: Start tacrolimus at 0.06 mg/kg PO BID. Day 0: Start MMF at 15 mg/kg PO b.i.d. from day 0 (PM dose only).

ELIGIBILITY:
Inclusion Criteria:

Patients with AML, ALL, CML, CLL, myelodysplastic syndrome (MDS), NHL, Hodgkin's disease (HD), or myeloma, who are at significantly higher than usual risk for mortality from conventional myeloablative allogeneic SCT due to age or comorbidities:

* Age ³ 50 years with AML or ALL in complete remission or with <10% blasts in bone marrow
* Age ³ 50 years with MDS or CML.
* Age > 50 years with lymphomas or myeloma, who have failed chemotherapy and are not candidates for an autologous transplant, or who have failed a prior autologous SCT.
* Patients of any age with CLL or low-grade NHL. Patients with CLL and low-grade NHL need to have failed at least first-line treatment, with an alkylating agent, fludarabine or 2-chlorodeoxyadenosine (2-CDA), or anti-CD20 monoclonal antibody rituximab.

  2. Patients with hematological malignancy relapsed after prior autologous transplantation.

  3. Patients at high-risk (>60%) of relapsing after autologous transplantation for hematological malignancies may receive allogeneic transplant as "consolidative immunotherapy". Diagnoses include multiple myeloma, non-Hodgkin's lymphoma, Hodgkin's lymphoma, AML, ALL and MDS. Minimal duration between autologous and allogeneic transplants is 4 weeks. 4. Patients of any age with hematologic malignancies treatable by allogeneic SCT, who, because of pre-existing medical conditions, are considered to be at significantly increased risk for transplant toxicity using high-dose transplant regimens. 5. Patients with metastatic renal cell carcinoma. Must have include good performance status (Karnofsky score > 60%), no active brain metastases, life expectancy > 6 months, absence of bulky liver metastases. Patients will be treated on other active disease-specific protocols when available. 6. Patients with other malignant diseases treatable with allogeneic SCT may be eligible for this protocol on a case by case basis, if approved by the principal investigator and the BMT attending physicians group. 7. Available HLA-identical sibling donor, or a phenotypically HLA-matched family member. 8. Age < 70 years.

Exclusion Criteria:

1. Patients with hematological malignancies eligible for a curative autologous SCT: intermediate- or high-grade NHL with chemo-sensitive first relapse. HD with chemo-sensitive first relapse.
2. Age <50 years and eligible for a conventional myeloablative allogeneic SCT.
3. Patients with rapidly progressive intermediate or high- grade NHL, unless in minimal disease state.
4. Patients with active uncontrolled CNS involvement with malignancy.
5. Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment.
6. Females who are pregnant.
7. Patients who are HIV positive
8. Organ dysfunction

   1. Left ventricle ejection fraction < 35%.
   2. DLCO <35% of predicted, or receiving continuous supplementary oxygen.
   3. Liver function tests: total bilirubin >2x the upper limit of normal, and/or transaminases >4x the upper limit of normal.
   4. Karnofsky score <50 for patients < 60 years, or <70 for patients aged 60 - 69 years (see appendix B).
   5. Creatinine clearance < 60 ml/min.
   6. Patients with hypertension that is poorly controlled on antihypertensive therapy.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-03

PRIMARY OUTCOMES:
The main endpoints are day 100 mortality and acute GVHD.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A McSweeney, MD, Principal Investigator — Colorado Blood Cancer Institute
Locations (1):
- Rocky Mountain Blood and Marrow Transplant Program, Denver, Colorado, United States